CLINICAL TRIAL: NCT03210428
Title: Quantitative MR Imaging in Locally Advanced Cervical Cancer Sub-study Under the EMBRACE II Protocol
Brief Title: Quantitative MR Imaging in Locally Advanced Cervical Cancer
Acronym: IQ-EMBRACE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Collaborators: The Netherlands Cancer Institute (Other)
Responsible Party: Principal Investigator, Jesper Kallehauge, Medical Physicist, Aarhus University Hospital
Other Study IDs: 57480
Record Dates: First submitted 2017-07-03; First posted 2017-07-07 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Neoplasms; Functional Magnetic Resonance Imaging; Radiotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypoxic tumour cells within the primary tumour have shown prognostic importance for local and metastatic disease control in several cancer sites. Radioresistant hypoxic cells diminish the rate of local control, and the hypoxia driven increase in metastatic potential of the tumour and lowers the rate of distant disease control. DCE MR imaging has been used to quantify the extent of poor perfusion regions within cervical tumours and it has been shown to be a surrogate of hypoxia. Furthermore, a number of studies have demonstrated that DCE MR is predictive of disease failure in cervix cancer.

The EMBRACE II study will implement an imaging sub-study, which will evaluate the value of quantitative MR imaging to identify patients at increased risk of disease recurrence (local, nodal and systemic).

DETAILED DESCRIPTION:
Radiotherapy is an important treatment modality in the management of cancers of the uterine cervix. About half of patients with cervical cancer receive definitive radiotherapy in the course of their disease. Radiotherapy is most often administered as a combination of external beam radiotherapy (EBRT) and brachytherapy (BT). In the late 90's a major breakthrough in cervical cancer radiotherapy took place with the introduction of MR image guidance of BT. By performing MR imaging before each BT implant it is possible adapt the dose given by BT to the anatomy of each individual patient taking into account not only the position of organs at risk (bladder, rectum and sigmoid) but also the tumour regression induced by the preceding EBRT and chemotherapy.

Functional imaging that reflects hypoxia, metabolism, heamodynamics and tissue structure have been applied to locally advanced cervical cancer with the goal to identify imaging markers that may predict outcome early on and improve tissue classification. DCE-MRI may be the most investigated so far for locally advanced cervical cancer. A comprehensive literature review including papers investigating the prognostic value of DCE-MRI in patients with locally advanced cervical cancer identified 20 papers from 10 research groups, with a median number of 30 patients (range 7-102 patients). A total number of 17 papers publish a positive association between pre-treatment DCE-MRI and outcome in terms of local control or disease free survival (1-17). However, not all studies present independent cohorts of patients. Three papers show no effect (18-20) The studies on cervical cancer points in the direction that DCE-MRI has the capability to identify aggressive forms of cervical cancer, and that the pre-treatment measurements may serve as, predictive markers for outcome after chemo-radiotherapy. The largest studies indicate that in particular the tumour fraction with the lowest signal enhancement is an important parameter, though the diversity in methodology is significant.

Diffusion weighted MRI (DWI-MRI) has to a lesser extent than DCE-MRI been investigated in locally advanced cervical cancer. Most studies using DWI-MRI in cervical cancer have investigated its diagnostic capabilities (21-28) all concluding high sensitivity and specificity (review by Kundu et al. (29)). The Toronto group; McVeight et al. (26) and later Gladwish et al. (30) found prior to the onset of treatment that the highest 90th % ADC value correlated with response, similar finding was found by the group in Tianjin; Liu et al. (22). Both groups found that higher ADC value insides the tumour was predictive of poor response to treatment and suggest the higher ADC to be connected to tumour necrosis. When tumour necrosis, occur there is loss of cell membrane integrity and therefore an increase in the extracellular volume and a decrease in intracellular volume effectively increasing the ADC. Conversely, the group from London UK; Harry et al. (31) and Somoye et al. (32) showed no correlation to treatment response at the time prior to treatment. Instead the ADC at 2 weeks (and the change in ADC) into treatment was predictive of treatment response and prognostic of patient outcome. Finally, Marconi et al. (33) found a relation between minimum ADC in the tumor and both DSS and DFS.

This is an observational prospective, non-randomized study in which patients with locally advanced cervical cancer included in the EMBRACE II study can enroll. The study will be carried out in 8-15 EMBRACE centres. MRI will be carried out prior to radiotherapy. The details of the MRI exams will differ from standard clinical practice in the centres, but will be consistent with international guidelines for cervix MRI. The exam will include T1, T2, diffusion, and dynamic contrast-enhanced imaging. At time of brachytherapy, the treatment planning MRI will additionally include DWI and qT2. Patients will be followed up according to the EMBRACE II follow-up schedule.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the EMBRACE study (see inclusion criteria in the EMBRACE protocol)
* Patients without previous record of allergic reaction to infusion of protocol related contrast media (Gadolinium-based)
* Patients with sufficient kidney function according to local regulations
* Patient informed consent

Exclusion Criteria:

* According to EMBRACE II protocol
* Patients with active infection or severe medical condition

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Yearly, each EMBRACE II centre is expected to enrol 10-20 patients. The inclusion for the imaging protocol in a given centre is expected to be 70% of patients enrolled in EMBRACE II. We expect that at least 8 institutions will enrol 10 patients per year, which will result in minimum 80 patients per year, and thereby at least 320 patients within the 4-year study period. This number is sufficient to meet the required number of patients for the hypotheses in the overall patient population (sample size 196 patients) and in the high-risk patients (sample size 248 patients )
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2018-10-18 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Disease control measure | 5 years
  To evaluate the sensitivity and specificity of dynamic contrast enhanced (DCE-MRI) to identify patients who have increased risk of disease recurrence (local, nodal, systemic) after radio-chemotherapy of cervix cancer

SECONDARY OUTCOMES:
Radiomics | 5 years
  To apply radiomics for identification of patients who have increased risk of disease recurrence (local, nodal, systemic) after radio-chemotherapy of cervix cancer. Radiomics analysis will include features from DCE-MRI, DWI and quantitative T2 imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Background] Mayr NA, Huang Z, Wang JZ, Lo SS, Fan JM, Grecula JC, Sammet S, Sammet CL, Jia G, Zhang J, Knopp MV, Yuh WT. Characterizing tumor heterogeneity with functional imaging and quantifying high-risk tumor volume for early prediction of treatment outcome: cervical cancer as a model. Int J Radiat Oncol Biol Phys. 2012 Jul 1;83(3):972-9. doi: 10.1016/j.ijrobp.2011.08.011. Epub 2011 Dec 28. PMID 22208967
- [Background] Mayr NA, Wang JZ, Zhang D, Grecula JC, Lo SS, Jaroura D, Montebello J, Zhang H, Li K, Lu L, Huang Z, Fowler JM, Wu DH, Knopp MV, Yuh WT. Longitudinal changes in tumor perfusion pattern during the radiation therapy course and its clinical impact in cervical cancer. Int J Radiat Oncol Biol Phys. 2010 Jun 1;77(2):502-8. doi: 10.1016/j.ijrobp.2009.04.084. Epub 2009 Sep 21. PMID 19775824
- [Background] Andersen EK, Hole KH, Lund KV, Sundfor K, Kristensen GB, Lyng H, Malinen E. Dynamic contrast-enhanced MRI of cervical cancers: temporal percentile screening of contrast enhancement identifies parameters for prediction of chemoradioresistance. Int J Radiat Oncol Biol Phys. 2012 Mar 1;82(3):e485-92. doi: 10.1016/j.ijrobp.2011.05.050. Epub 2011 Oct 17. PMID 22014954
- [Background] Loncaster JA, Carrington BM, Sykes JR, Jones AP, Todd SM, Cooper R, Buckley DL, Davidson SE, Logue JP, Hunter RD, West CM. Prediction of radiotherapy outcome using dynamic contrast enhanced MRI of carcinoma of the cervix. Int J Radiat Oncol Biol Phys. 2002 Nov 1;54(3):759-67. doi: 10.1016/s0360-3016(02)02972-3. PMID 12377328
- [Background] Takayama Y, Ohno T, Kishimoto R, Kato S, Yoneyama R, Kandatsu S, Tsujii H, Obata T. Prediction of early response to radiotherapy of uterine carcinoma with dynamic contrast-enhanced MR imaging using pixel analysis of MR perfusion imaging. Magn Reson Imaging. 2009 Apr;27(3):370-6. doi: 10.1016/j.mri.2008.07.007. Epub 2008 Sep 2. PMID 18768283
- [Background] Semple SI, Harry VN, Parkin DE, Gilbert FJ. A combined pharmacokinetic and radiologic assessment of dynamic contrast-enhanced magnetic resonance imaging predicts response to chemoradiation in locally advanced cervical cancer. Int J Radiat Oncol Biol Phys. 2009 Oct 1;75(2):611-7. doi: 10.1016/j.ijrobp.2009.04.069. PMID 19735887
- [Background] Mayr NA, Yuh WT, Zheng J, Ehrhardt JC, Magnotta VA, Sorosky JI, Pelsang RE, Oberley LW, Hussey DH. Prediction of tumor control in patients with cervical cancer: analysis of combined volume and dynamic enhancement pattern by MR imaging. AJR Am J Roentgenol. 1998 Jan;170(1):177-82. doi: 10.2214/ajr.170.1.9423627.
- [Background] Mayr NA, Yuh WT, Magnotta VA, Ehrhardt JC, Wheeler JA, Sorosky JI, Davis CS, Wen BC, Martin DD, Pelsang RE, Buller RE, Oberley LW, Mellenberg DE, Hussey DH. Tumor perfusion studies using fast magnetic resonance imaging technique in advanced cervical cancer: a new noninvasive predictive assay. Int J Radiat Oncol Biol Phys. 1996 Oct 1;36(3):623-33. doi: 10.1016/s0360-3016(97)85090-0. PMID 8948347
- [Background] Mayr NA, Yuh WT, Arnholt JC, Ehrhardt JC, Sorosky JI, Magnotta VA, Berbaum KS, Zhen W, Paulino AC, Oberley LW, Sood AK, Buatti JM. Pixel analysis of MR perfusion imaging in predicting radiation therapy outcome in cervical cancer. J Magn Reson Imaging. 2000 Dec;12(6):1027-33. doi: 10.1002/1522-2586(200012)12:63.0.co;2-5. PMID 11105046
- [Background] Mannelli L, Patterson AJ, Zahra M, Priest AN, Graves MJ, Lomas DJ, Tan LT, Crawford R, Brenton J, Sala E. Evaluation of nonenhancing tumor fraction assessed by dynamic contrast-enhanced MRI subtraction as a predictor of decrease in tumor volume in response to chemoradiotherapy in advanced cervical cancer. AJR Am J Roentgenol. 2010 Aug;195(2):524-7. doi: 10.2214/AJR.09.3437. PMID 20651213
- [Background] Zahra MA, Tan LT, Priest AN, Graves MJ, Arends M, Crawford RA, Brenton JD, Lomas DJ, Sala E. Semiquantitative and quantitative dynamic contrast-enhanced magnetic resonance imaging measurements predict radiation response in cervix cancer. Int J Radiat Oncol Biol Phys. 2009 Jul 1;74(3):766-73. doi: 10.1016/j.ijrobp.2008.08.023. Epub 2008 Nov 18. PMID 19019563
- [Background] Gong QY, Brunt JN, Romaniuk CS, Oakley JP, Tan LT, Roberts N, Whitehouse GH, Jones B. Contrast enhanced dynamic MRI of cervical carcinoma during radiotherapy: early prediction of tumour regression rate. Br J Radiol. 1999 Dec;72(864):1177-84. doi: 10.1259/bjr.72.864.10703475.
- [Background] Andersen EK, Kristensen GB, Lyng H, Malinen E. Pharmacokinetic analysis and k-means clustering of DCEMR images for radiotherapy outcome prediction of advanced cervical cancers. Acta Oncol. 2011 Aug;50(6):859-65. doi: 10.3109/0284186X.2011.578586. PMID 21767185
- [Background] Mayr NA, Wang JZ, Zhang D, Montebello JF, Grecula JC, Lo SS, Fowler JM, Yuh WT. Synergistic effects of hemoglobin and tumor perfusion on tumor control and survival in cervical cancer. Int J Radiat Oncol Biol Phys. 2009 Aug 1;74(5):1513-21. doi: 10.1016/j.ijrobp.2008.09.050. Epub 2009 Mar 13. PMID 19286329
- [Background] Huang Z, Yuh KA, Lo SS, Grecula JC, Sammet S, Sammet CL, Jia G, Knopp MV, Wu Q, Beauchamp NJ 3rd, Yuh WT, Wang R, Mayr NA. Validation of optimal DCE-MRI perfusion threshold to classify at-risk tumor imaging voxels in heterogeneous cervical cancer for outcome prediction. Magn Reson Imaging. 2014 Dec;32(10):1198-205. doi: 10.1016/j.mri.2014.08.039. Epub 2014 Aug 29. PMID 25179141
- [Background] Torheim T, Malinen E, Kvaal K, Lyng H, Indahl UG, Andersen EK, Futsaether CM. Classification of dynamic contrast enhanced MR images of cervical cancers using texture analysis and support vector machines. IEEE Trans Med Imaging. 2014 Aug;33(8):1648-56. doi: 10.1109/TMI.2014.2321024. Epub 2014 Apr 29. PMID 24802069
- [Background] Donaldson SB, Buckley DL, O'Connor JP, Davidson SE, Carrington BM, Jones AP, West CM. Enhancing fraction measured using dynamic contrast-enhanced MRI predicts disease-free survival in patients with carcinoma of the cervix. Br J Cancer. 2010 Jan 5;102(1):23-6. doi: 10.1038/sj.bjc.6605415. Epub 2009 Nov 17. PMID 19920831
- [Background] Mayr NA, Yuh WT, Jajoura D, Wang JZ, Lo SS, Montebello JF, Porter K, Zhang D, McMeekin DS, Buatti JM. Ultra-early predictive assay for treatment failure using functional magnetic resonance imaging and clinical prognostic parameters in cervical cancer. Cancer. 2010 Feb 15;116(4):903-12. doi: 10.1002/cncr.24822. PMID 20052727
- [Background] Kim JH, Kim CK, Park BK, Park SY, Huh SJ, Kim B. Dynamic contrast-enhanced 3-T MR imaging in cervical cancer before and after concurrent chemoradiotherapy. Eur Radiol. 2012 Nov;22(11):2533-9. doi: 10.1007/s00330-012-2504-4. Epub 2012 Jun 1. PMID 22653283
- [Background] Boss EA, Massuger LF, Pop LA, Verhoef LC, Huisman HJ, Boonstra H, Barentsz JO. Post-radiotherapy contrast enhancement changes in fast dynamic MRI of cervical carcinoma. J Magn Reson Imaging. 2001 Apr;13(4):600-6. doi: 10.1002/jmri.1084. PMID 11276105
- [Background] Chen YB, Hu CM, Chen GL, Hu D, Liao J. Staging of uterine cervical carcinoma: whole-body diffusion-weighted magnetic resonance imaging. Abdom Imaging. 2011 Oct;36(5):619-26. doi: 10.1007/s00261-010-9642-4. PMID 20730423
- [Background] Liu Y, Bai R, Sun H, Liu H, Wang D. Diffusion-weighted magnetic resonance imaging of uterine cervical cancer. J Comput Assist Tomogr. 2009 Nov-Dec;33(6):858-62. doi: 10.1097/RCT.0b013e31819e93af. PMID 19940650
- [Background] Naganawa S, Sato C, Kumada H, Ishigaki T, Miura S, Takizawa O. Apparent diffusion coefficient in cervical cancer of the uterus: comparison with the normal uterine cervix. Eur Radiol. 2005 Jan;15(1):71-8. doi: 10.1007/s00330-004-2529-4. Epub 2004 Nov 5. PMID 15538578
- [Background] Kilickesmez O, Bayramoglu S, Inci E, Cimilli T, Kayhan A. Quantitative diffusion-weighted magnetic resonance imaging of normal and diseased uterine zones. Acta Radiol. 2009 Apr;50(3):340-7. doi: 10.1080/02841850902735858. PMID 19235579
- [Background] Charles-Edwards EM, Messiou C, Morgan VA, De Silva SS, McWhinney NA, Katesmark M, Attygalle AD, DeSouza NM. Diffusion-weighted imaging in cervical cancer with an endovaginal technique: potential value for improving tumor detection in stage Ia and Ib1 disease. Radiology. 2008 Nov;249(2):541-50. doi: 10.1148/radiol.2491072165. PMID 18936313
- [Background] McVeigh PZ, Syed AM, Milosevic M, Fyles A, Haider MA. Diffusion-weighted MRI in cervical cancer. Eur Radiol. 2008 May;18(5):1058-64. doi: 10.1007/s00330-007-0843-3. Epub 2008 Jan 12. PMID 18193428
- [Background] Xue HD, Li S, Sun F, Sun HY, Jin ZY, Yang JX, Yu M. Clinical application of body diffusion weighted MR imaging in the diagnosis and preoperative N staging of cervical cancer. Chin Med Sci J. 2008 Sep;23(3):133-7. doi: 10.1016/s1001-9294(09)60027-4. PMID 18853846
- [Background] Hoogendam JP, Klerkx WM, de Kort GA, Bipat S, Zweemer RP, Sie-Go DM, Verheijen RH, Mali WP, Veldhuis WB. The influence of the b-value combination on apparent diffusion coefficient based differentiation between malignant and benign tissue in cervical cancer. J Magn Reson Imaging. 2010 Aug;32(2):376-82. doi: 10.1002/jmri.22236. PMID 20677265
- [Background] Kundu S, Chopra S, Verma A, Mahantshetty U, Engineer R, Shrivastava SK. Functional magnetic resonance imaging in cervical cancer: current evidence and future directions. J Cancer Res Ther. 2012 Jan-Mar;8(1):11-8. doi: 10.4103/0973-1482.95167. PMID 22531506
- [Background] Gladwish A, Milosevic M, Fyles A, Xie J, Halankar J, Metser U, Jiang H, Becker N, Levin W, Manchul L, Foltz W, Han K. Association of Apparent Diffusion Coefficient with Disease Recurrence in Patients with Locally Advanced Cervical Cancer Treated with Radical Chemotherapy and Radiation Therapy. Radiology. 2016 Apr;279(1):158-66. doi: 10.1148/radiol.2015150400. Epub 2015 Oct 27. PMID 26505922
- [Background] Harry VN, Semple SI, Gilbert FJ, Parkin DE. Diffusion-weighted magnetic resonance imaging in the early detection of response to chemoradiation in cervical cancer. Gynecol Oncol. 2008 Nov;111(2):213-20. doi: 10.1016/j.ygyno.2008.07.048. Epub 2008 Sep 6. PMID 18774597
- [Background] Somoye G, Harry V, Semple S, Plataniotis G, Scott N, Gilbert FJ, Parkin D. Early diffusion weighted magnetic resonance imaging can predict survival in women with locally advanced cancer of the cervix treated with combined chemo-radiation. Eur Radiol. 2012 Nov;22(11):2319-27. doi: 10.1007/s00330-012-2496-0. Epub 2012 Jun 1. PMID 22653281
- [Background] Marconi DG, Fregnani JH, Rossini RR, Netto AK, Lucchesi FR, Tsunoda AT, Kamrava M. Pre-treatment MRI minimum apparent diffusion coefficient value is a potential prognostic imaging biomarker in cervical cancer patients treated with definitive chemoradiation. BMC Cancer. 2016 Jul 28;16:556. doi: 10.1186/s12885-016-2619-0. PMID 27469349
- See also: EMBRACE study webpage — https://www.embracestudy.dk/